CLINICAL TRIAL: NCT00365404
Title: Weight Management, Physical Activity, Less Disability in Rheumatoid and Osteoarthritis
Brief Title: Activity, Rheumatoid and Osteoarthritis, and Weight Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single
Other Study IDs: 01802-03-C; R04/CCR523273-03-2
Record Dates: First submitted 2006-08-16; First posted 2006-08-17 (Estimated); Last update posted 2015-11-26 (Estimated); Status verified 2006-07

CONDITIONS: Rheumatoid Arthritis; Osteoarthritis
Keywords: Behavioral change; Weight management; Physical activity
MeSH Terms: conditions — Arthritis, Rheumatoid; Osteoarthritis; Motor Activity | interventions — Diet

INTERVENTIONS:
Behavioral: Diet and exercise promotion

SUMMARY:
The purpose of the study was to implement well-developed guidelines for arthritis management beyond acute medical management to independent community living by modifying existing weight management and physical activity promotion programs for people with disabling arthritis.

Our hypotheses were:

1. Existing individual, health care system, and community strategies to promote physical activity and weight management can effectively be modified and expanded to include those with debilitating joint diseases.
2. People with inflammatory joint disease can have healthy physical activity levels and weight at home and in the community.
3. The effect of these interventions will be higher quality of life, lower depression rates, modest pain levels, and functional independence.

DETAILED DESCRIPTION:
Park Nicollet Clinic and the Institute for Clinical Systems Integration have spent several million dollars developing evidence-based care guidelines and intervention strategies for a wide range of common illnesses. Included in the degenerative joint disease guideline are recommendations for the management of two inter-related risk factors for increased disability: obesity and lack of physical activity. This application seeks to integrate disability prevention programs into the post-acute management of rheumatoid and osteoarthritis.

Our specific aims are to: (1) Modify well-established weight management techniques and physical activity promotion interventions according to Institute for Clinical Systems Integration recommendations for use by the broader community of individuals with potentially disabling rheumatoid and osteoarthritis; (2) Implement these interventions within a diverse patient population identified within an integrated health care system; (3) Demonstrate the short and long term impact of these interventions on patients suffering from debilitating joint disease; and (4) Facilitate incorporation of these interventions by other communities and clinical settings to enhance the longer-term well being of those with disabilities.

To achieve our aims, we will modify existing weight management and physical activity promotion strategies across the continuum of care. Through patient focus groups, a clinical advisory board, a community advisory board, and pilot testing, key stakeholders will help assure effective program design and implementation strategies as well as development of sustainable interventions. Using pre- and post-intervention surveys and simple measures of physical ability and weight, we will demonstrate the effect of these interventions on physical activity levels and weight; assess the effect of the interventions on pain, quality of life, depression, and functional capacity in those diagnosed with rheumatoid or osteoarthritis; and document the implementation strategies for the community interventions.

Our aims and hypotheses are consistent with the overarching goals of Healthy People 2010: (1) to increase quality and years of healthy life and (2) to eliminate health disparities. We address two focus areas, (2) arthritis and (6) disability and secondary conditions. Our intervention targets two of the leading health indicators: physical activity and overweight and obesity.

ELIGIBILITY:
Inclusion Criteria:

* Adult men and women
* A medical visit at one of six Park Nicollet Health System sites from November 2003 through June 2004.
* ICD-9 visit code of 714.0, 715.90 or 715.95 through 715.97
* Patient's clinician provided written consent to invite participation
* Patients had previously consented to be contacted for research purposes.

Exclusion Criteria:

* The patient was unaware of a medical diagnosis of arthritis.
* They did not report having a medical provider they could call with arthritis-related questions
* Arthritis-related problems for less than nine months duration for rheumatoid arthritis, less than three months for osteoarthritis.
* Scheduled for surgery.
* History of lower extremity joint replacement.
* Less than daily arthritis pain or problems.
* History of chest pain or medically restricted activity.
* Unable to participate for 12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 465
Dates: Start 2003-10; Study Completion 2006-02

PRIMARY OUTCOMES:
Normal body mass index is normal
At least four days of 20 minutes exercise in past seven

SECONDARY OUTCOMES:
Weight loss of five pounds
Increased exercise days by 2
Improved quality of life (including reduced pain) as measured with the AIMS-2
Improved dietary characteristics as measured with the Block FFQ
Increased physical activity as measured with the Physical ACtivity History
Reduced depressive symptoms via CES-D
Improved physical performance

CONTACTS AND LOCATIONS:
Overall Officials: Barbara L Braun, PhD, Principal Investigator — HealthPartners Institute
Locations (1):
- Park Nicollet Institute, Saint Louis Park, Minnesota, United States